CLINICAL TRIAL: NCT02330588
Title: Working With Parents to Prevent Childhood Obesity: A Primary Care-based Study
Brief Title: The Resource Information Program for Parents on Lifestyle and Education
Acronym: RIPPLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RIPPLE-0613
Record Dates: First submitted 2014-12-17; First posted 2015-01-05 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Pediatric Obesity
Keywords: Obesity; Prevention; Pediatric; Parents; Primary Care; eHealth; Internet
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Eat It! (Injunctive Feedback) (Experimental): Parents are presented with two questions about portion size and sugar-sweetened beverages; answers are contrasted with injunctive feedback (i.e., Canadian guidelines).
  Interventions: Behavioral: Eat It
- Eat It! (Normative Feedback) (Experimental): Parents are presented with two questions about portion size and sugar-sweetened beverages; answers are contrasted with normative feedback (i.e., referent data from Canadian children).
  Interventions: Behavioral: Eat It
- Move It! (Injunctive Feedback) (Experimental): Parents are presented with two questions about screen time and moderate-to-vigorous physical activity (MVPA); answers are contrasted with injunctive feedback (i.e., Canadian guidelines).
  Interventions: Behavioral: Move It
- Move It! (Normative Feedback) (Experimental): Parents are presented with two questions about screen time and moderate-to-vigorous physical activity (MVPA); answers are contrasted with normative feedback (i.e., referent data from Canadian children).
  Interventions: Behavioral: Move It
- eHealth Control (Placebo Comparator): Parents randomly assigned to the control arm will include information on children's lifestyle behaviors only (no intervention questions).
  Interventions: Behavioral: eHealth Control

INTERVENTIONS:
Behavioral: Eat It — The SBIRT (Screening, Brief Intervention, Referral to Treatment), called RIPPLE (Resource Information Program for Parents on Lifestyle Education) was delivered on a study-designated tablet and designed to (1) screen children's weight status, (2) deliver a brief intervention*, and (3) provide parents with the opportunity select resources and services to help prevent obesity in children.
  *Two brief questions about children's grain portion sizes and sugar sweetened beverage intake were presented.
  Arms: Eat It! (Injunctive Feedback); Eat It! (Normative Feedback)
Behavioral: Move It — The SBIRT (Screening, Brief Intervention, Referral to Treatment), called RIPPLE (Resource Information Program for Parents on Lifestyle Education) was delivered on a study-designated tablet and designed to (1) screen children's weight status, (2) deliver a brief intervention*, and (3) provide parents with the opportunity select resources and services to help prevent obesity in children.
  *Two brief questions about children's moderate-to-vigorous physical activity (MVPA) and screen time were presented.
  Arms: Move It! (Injunctive Feedback); Move It! (Normative Feedback)
Behavioral: eHealth Control — The eHealth Control group (1) screened children's weight status, and (2) provided parents with the opportunity select resources and services to help prevent obesity in children.
  Other Names: Heads Up
  Arms: eHealth Control

SUMMARY:
Childhood obesity is an urgent public health issue. Roughly one-quarter of Canadian children are overweight, putting them at risk for chronic diseases. Because most families access health services in primary care, it is an ideal venue for obesity prevention. Specifically, programs in primary care can prevent unhealthy weight gain in healthy weight children (primary prevention) AND reduce unhealthy weight gain in children who are already overweight (secondary prevention). Parents play a key role in children's health, so it is vital to include parents in strategies to prevent childhood obesity.

The following objectives of this study are to: (i) develop a web-based, brief program for parents as an educational tool to motivate parents to support healthy lifestyles in children, and access community resources and health services that can prevent childhood obesity; (ii) assess the acceptability of the program using focus groups with parents, and pediatric-focused health care professionals, trainees, and administrators; and (iii) recruit parents (n=200) in primary care and collect data at baseline and 1-month follow-up to explore if the program led to changes in parents' motivation to support their children's lifestyle habits, and families' use of resources and health services to prevent childhood obesity.

It is hypothesized that the developed screening, brief intervention, and referral to treatment (SBIRT) will (i) encourage parents of healthy weight children to seek resources to eat healthfully and be physically active to maintain their weight status (primary [1°] prevention), and (ii) guide parents of unhealthy weight children to access educational tools and community services to reduce their child's obesity and associated health risks (secondary [2°] prevention).

By providing families with tailored feedback, practical educational tools, and information on local health services, this research will help to address oft-cited barriers primary care clinicians commonly report when providing effective obesity-related health services, and encourage family self-management of obesity-related behaviors.

DETAILED DESCRIPTION:
Background: There is urgent need to develop and evaluate innovative, evidence-based, and sustainable approaches for pediatric obesity in accessible settings. One such approach, the screening, brief intervention, and referral to treatment (SBIRT), has been used to address preventable health concerns, such as hazardous drinking; this time- and resource-limited approach delivers a brief, theoretically-driven intervention to increase awareness of a health concern and provides the respondent with feedback and information on relevant resources. This approach is suited to obesity prevention as it can enhance parents' awareness and concern for children's lifestyle behaviors, remove social barriers and provide anonymity for families, and overcome limited availability of obesity-related health services.

Setting. This study will take place at a centrally-located Edmonton pediatric clinic housed within the Edmonton Oliver Primary Care Network (EOPCN). Primary care (PC) represents an accessible, relevant, and appropriate venue to prevent pediatric obesity because (i) PC often represents families' first point of contact with the health care system, (ii) the goals and priorities of PC clinics are well-aligned with primary and secondary prevention of chronic diseases, and (iii) patients typically access health care services throughout the life course, therefore representing a suitable environment to capture longitudinal data.

Phase I. The objective of this phase is to develop a web-based, theoretically-driven SBIRT to enhance parents' awareness, concern for, and motivation to support children's lifestyle behaviors. The SBIRT (RIPPLE; the Resource Information Program for Parents on Lifestyle and Education) will screen children of all weight statuses, deliver a brief intervention regarding children's lifestyle behaviors to parents, and provide parents with a menu of resources and community resources to facilitate the prevention of obesity in children. The intervention has been informed by the Norm Activation Model, and a survey following the intervention will test psychosocial constructs from the Theory of Planned Behavior and Health Belief Model. Parents will receive a personalized report based on their intervention responses and selected resources and services; parents will have the option to email this report to themselves.

Phase II. The objective of this phase is to refine the SBIRT using focus groups. Participants (n=30) will include parents, and pediatric-focused administrators, health care providers, research coordinators, and graduate trainees. Focus groups will query participants' overall perceptions of the program; specifically, impressions regarding likability, acceptability, satisfaction, and feasibility of incorporating the intervention into clinical practice. Focus group discussions will be transcribed in real-time using a court reporter, which will optimize transcription accuracy and ensure confidentiality. The method of Qualitative Description (QD) will be used to develop a rich and explicit description of the phenomena. QD necessitates less interpretive interference on behalf of the researcher, therefore representing an accurate and realistic embodiment of participants' discussion.

Phase III (RCT). The objective of this phase is to recruit parents (n=200) from a pediatric primary care clinic to enroll in the RCT. This double-blinded, parallel-design RCT will adhere to CONSORT guidelines. The allocation sequence will be electronically generated and blocked randomization (5 arms; block size of five) will be used to ensure equal group sizes throughout the study. Research assistants will be blinded to participants' intervention assignment and participants will not be aware if they have received the intervention or control.

Parents will be eligible for the study if they speak and read English, and have a 5 - 17 year old child who is present at the appointment with a non-urgent medical issue. Data will be collected at (i) baseline during delivery of the online RCT and (ii) 1-month follow-up to assess time-related changes in parents' psychosocial constructs (e.g., intention to change children's lifestyle behaviors; primary outcome) and families' utilization of resources and health services to facilitate healthy lifestyle behaviors (secondary outcome). Follow-up will include email delivery of a survey measure identical to that administered at baseline. Given rates of attrition tend to increase over time parents' access to the online personalized report will serve as a proxy of participation if the online survey is not completed.

Continuous variables will be described by univariate summaries; frequency distributions will be determined for categorical variables. Participant characteristics (e.g., weight status, child sex) will be examined to assess equivalence of intervention groups at baseline, and attrition tendencies across sub-groups will be examined using two-way ANOVA. Multilevel modelling will be used to assess intra- and inter-level individual and group change in the primary and secondary outcomes; this form of analysis is appropriate when observations are nested within groups and/or multiple time points. Estimates of effect sizes will be based on percent change in primary outcomes. Significance will be p<0.05.

Significance & Future Directions. The SBIRT is designed to encourage self-management by providing families with tailored feedback and linking them with appropriate and relevant resources to facilitate children's healthy lifestyle behaviors. Findings from this study will inform future intervention refinement and implementation into everyday clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* parents of children 5-17 years of age
* parents speak and read English

Exclusion Criteria:

* children present with urgent medical issues (e.g., febrile, acute asthma attack)
* children attend appointment without legal guardian
* parents do not have sufficient time (15-20 minutes) to complete the intervention

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoff DC Ball, PhD, Principal Investigator — University of Alberta
Locations (1):
- The Allin Clinic, Edmonton Oliver Primary Care Network, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Campbell M, Benton JM, Werk LN. Parent perceptions to promote a healthier lifestyle for their obese child. Soc Work Health Care. 2011;50(10):787-800. doi: 10.1080/00981389.2011.597316. PMID 22136345
- [Derived] Avis JL, Cave AL, Donaldson S, Ellendt C, Holt NL, Jelinski S, Martz P, Maximova K, Padwal R, Wild TC, Ball GD. Working With Parents to Prevent Childhood Obesity: Protocol for a Primary Care-Based eHealth Study. JMIR Res Protoc. 2015 Mar 25;4(1):e35. doi: 10.2196/resprot.4147. PMID 25831265
- See also: Study-dedicated blog to provide updates and news to research team — http://rippleprogram.wordpress.com/
- See also: RCT publication (Byrne et al., 2016; Pediatric Obesity) — http://onlinelibrary.wiley.com/doi/10.1111/ijpo.12200/abstract

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 226 participants were recruited from July to October 2015 in a pediatric primary care clinic (Figure 1; http://onlinelibrary.wiley.com/doi/10.1111/ijpo.12200/abstract).
Groups:
- Eat It (Injunctive Feedback): Parents are presented with two questions about portion size and sugar-sweetened beverages; answers are contrasted with injunctive feedback (i.e., Canadian guidelines).
- Eat It (Normative Feedback): Parents are presented with two questions about portion size and sugar-sweetened beverages; answers are contrasted with normative feedback (i.e., referent data from Canadian children).
- Move It (Injunctive Feedback): Parents are presented with two questions about screen time and moderate-to-vigorous physical activity (MVPA); answers are contrasted with injunctive feedback (i.e., Canadian guidelines).
- Move It (Normative Feedback): Parents are presented with two questions about screen time and moderate-to-vigorous physical activity (MVPA); answers are contrasted with normative feedback (i.e., referent data from Canadian children).
Period: Overall Study
Arm/Group | Eat It (Injunctive Feedback) | Eat It (Normative Feedback) | Move It (Injunctive Feedback) | Move It (Normative Feedback) | eHealth Control
Started | 44 | 43 | 46 | 46 | 47
Completed | 28 | 25 | 31 | 24 | 28
Not Completed | 16 | 18 | 15 | 22 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm (Eat It, Injunctive Feedback) | Intervention Arm (Eat It, Normative Feedback) | Intervention Arm (Move It, Injunctive Feedback) | Intervention Arm (Move It, Normative Feedback) | eHealth Control Arm (Heads Up) | Total
Number analyzed (Participants) | 44 | 43 | 46 | 46 | 47 | 226
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 44 | 43 | 46 | 46 | 47 | 226
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (3.6) | 9.7 (3.2) | 10.3 (3.9) | 9.6 (3.5) | 10.2 (2.9) | 9.9 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 16 | 21 | 30 | 111
  Male | 20 | 23 | 30 | 25 | 17 | 115

OUTCOME MEASURES:

1. Primary Outcome: Feasibility (Parents' Interest in the SBIRT.)
Description: Parents' interest was determined by the proportion (indicated as a percentage) of parents that (i) enrolled among those approached to participate, (ii) 'opted in' to receive the tailored email report, and (iii) self-selected resources from the SBIRT; the latter two were recorded by back-end programming of the SBIRT.
Time Frame: Baseline
Population: Parents who participated at baseline.
Measure: Number; unit: percentage of parents
Groups:
- All Groups (Total): All groups (four brief interventions + eHealth control)
Arm/Group | All Groups (Total) | Eat It (Injunctive Feedback) | Eat It (Normative Feedback) | Move It (Injunctive Feedback) | Move It (Normative Feedback) | eHealth Control
Number analyzed (Participants) | 226 | 44 | 43 | 46 | 46 | 47
percentage of parents
  Proportion that Enrolled (%) | 84.3 | NA — Because enrollment happened prior to randomization, per-arm proportions are not available for proportion enrolled. | NA — Because enrollment happened prior to randomization, per-arm proportions are not available for proportion enrolled. | NA — Because enrollment happened prior to randomization, per-arm proportions are not available for proportion enrolled. | NA — Because enrollment happened prior to randomization, per-arm proportions are not available for proportion enrolled. | NA — Because enrollment happened prior to randomization, per-arm proportions are not available for proportion enrolled.
  Proportion that Opted into Tailored Report (%) | 63.7 | 61.4 | 62.3 | 78.2 | 52.2 | 63.8
  Proportion that Self-selected Resources (%) | 85.8 | 84.1 | 86.0 | 82.3 | 78.3 | 95.7

2. Primary Outcome: Feasibility (Parents' Uptake of the SBIRT)
Description: Parents' uptake was determined by parents' use (actual and self-reported) of obesity prevention resources (i.e., the proportion [reported in percentage] that actually or self-reported using resources out of the total number of participants that participated in follow-up), and the proportion (reported in percentage) of parents that reported discussing children's weight with their pediatrician immediately following the SBIRT.
Time Frame: One-month follow-up
Population: Participants who completed one-month follow-up.
Measure: Number; unit: percentage of participants
Groups:
- Feasibility (Uptake): All groups (brief intervention + eHealth control)
Arm/Group | Feasibility (Uptake) | Eat It (Injunctive Feedback) | Eat It (Normative Feedback) | Move It (Injunctive Feedback) | Move It (Normative Feedback) | eHealth Control
Number analyzed (Participants) | 136 | 28 | 25 | 31 | 24 | 28
percentage of participants
  Proportion Self-reported Use of Resources (%) | 41.2 | 35.7 | 36.0 | 45.2 | 37.5 | 46.4
  Proportion Actual use of Resources (%) | 16.0 | 25.0 | 8.0 | 16.1 | 16.7 | 17.9
  Proportion Reporting Discussing Weight with MD (%) | 52.2 | 35.7 | 40.0 | 58.1 | 50.0 | 46.4

3. Secondary Outcome: Parents' Concern About Children's Weight Status and Motivation to Change Lifestyle Behaviors Immediately Following the SBIRT.
Description: A brief, eight-item Likert scale questionnaire with established face validity has been adopted from Campbell et al. (2011) and will assess parents' concern for and motivation to support their child's lifestyle behaviors. Concern and motivation to change were measured on a 5-point Likert scale ('strongly disagree' [0] to 'strongly agree' [4]); for example, "I am ready to change my child's lifestyle behaviors", a 0 would indicate that participants strongly disagree with this statement.
Time Frame: Measured at baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale (0 to 4 Likert Scale)
Arm/Group | Eat It (Injunctive Feedback) | Eat It (Normative Feedback) | Move It (Injunctive Feedback) | Move It (Normative Feedback) | Heads Up (eHealth Control) | All Groups (Total)
Number analyzed (Participants) | 44 | 43 | 46 | 46 | 47 | 226
units on a scale (0 to 4 Likert Scale)
  Concern about Weight Status | 1.18 [0.73 to 1.64] | 0.88 [0.50 to 1.26] | 0.59 [0.26 to 0.91] | 0.52 [0.22 to 0.82] | 0.55 [0.27 to 0.83] | 0.74 [0.58 to 0.89]
  Motivation to Change Children's Lifestyle Behavior | 2.43 [2.01 to 2.85] | 2.28 [1.86 to 2.70] | 2.48 [2.06 to 2.89] | 2.70 [2.32 to 3.07] | 2.71 [2.43 to 3.00] | 2.52 [2.36 to 2.69]

ADVERSE EVENTS:
Arm/Group | Eat It (Injunctive) | Eat It (Normative) | Move It (Injunctive) | Move It (Normative) | eHealth Control
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/43 | 0/46 | 0/46 | 0/47
Other Adverse Events (participants affected / at risk) | 0/44 | 0/43 | 0/46 | 0/46 | 0/47

LIMITATIONS AND CAVEATS:
(1) The SBIRT did not include data collection of parents' self-reported concern and intention pre- and post-intervention, and (2) the study was developmental in nature and was not sufficiently powered to detect group differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No